CLINICAL TRIAL: NCT05555303
Title: Preventing Acquired Resistance: Strengthen TB Treatment by Adding Amikacin in the First Treatment Week of Multidrug-resistant Tuberculosis (Stake) Amendment to Study Protocol: "All-oral Shorter Treatment Regimen for Multidrug- and Rifampicin-resistant Tuberculosis (MDR/RR-TB): Evaluating Its Effectiveness, Safety and Impact on the Quality of Life of Patients in Rwanda" (ShORRT)
Brief Title: Preventing Acquired Resistance: Strengthen TB Treatment by Adding Amikacin in the First Treatment Week of Multidrug-resistant Tuberculosis
Acronym: Stake
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rwanda Biomedical Centre (Other)
Collaborators: Institute of Tropical Medicine (Other Government); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBC/RIDS012022
Record Dates: First submitted 2022-09-16; First posted 2022-09-26 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: multidrug- and rifampicin-resistant tuberculosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amikacin (Other)
  Interventions: Drug: Amikacin

INTERVENTIONS:
Drug: Amikacin — In addition to the all-oral RR-TB treatment, add two intramuscular doses each consisting of 30 mg amikacin/kg, a first dose on day 1 and a second dose on day 4, all in the first week of treatment.
  The amikacin solution will be admixed with a lidocaine solution in the syringe before administration.

SUMMARY:
Acquired drug-resistance is a major challenge for tuberculosis (TB) care programs. The 2020 WHO guidelines recommends replacing second-line injectables by bedaquiline in rifampicin-resistant TB (RR-TB) treatment regimens. However, recent reports show too high rates of acquired bedaquiline resistance. This may be explained by the delayed onset of action of bedaquiline. The investigators will study whether high-dose amikacin (a second-line injectable), administered during the first week of RR-TB treatment, is safe in 20 patients treated for RR-TB in Rwanda. If safe, further studies will assess whether adding amikacin in the first treatment week protect against acquired bedaquiline resistance. This study is embedded in an ongoing "Master study" of the ShORRT (short oral RR-TB) treatment regimen in Rwanda, a before/after study, with a retrospective cohort (before; the previously recommended second-line injectable-containing RR-TB regimen) and a prospective cohort (after: the newly recommended ShORRT regimen).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Master SHORRT study
* Able and willing to provide written informed consent for the present substudy "Stake"

Exclusion Criteria:

* Any audiometry abnormality (grade 1 or higher) on baseline audiometry
* History of kidney disease or baseline creatinine clearance below or equal to 60ml/min
* Pregnant or breastfeeding women
* History of previous injectable based tuberculosis treatment (including with streptomycin)
* < 18 years and > 65 years old
* Patient on NSAID or on diuretics

Master ShORRT study

Inclusion criteria:

* Is willing and able to give informed consent to be enrolled in the research project and for follow-up
* Has bacteriologically or molecularly confirmed TB with evidence of resistance to at least rifampicin

Exclusion criteria:

* Is unable to take oral medication;
* Must take any medications contraindicated with the medicines in the MDR/RR-TB regimen;
* Has a known allergy to any of the drugs in the MDR/RR-TB regimen;
* Has a QTcF interval of ≥ 500 msec; at baseline that does not correct with medical management.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
grade 3-4 AE likely or definitively related to amikacin | After 2 weeks of treatment
  Assess whether less than 14% of patients treated with the amikacin-strengthened regimen will experience a grade 3-4 adverse event likely or definitively related to the use of amikacin

SECONDARY OUTCOMES:
turnaround times | at the end of treatment week 2 (+/- 3 d)
  Assess the turnaround times to inform the feasibility of doing the tests proposed in this study for the assessment of the response to the use of two doses of amikacin
testing coverage | at the end of treatment week 2 (+/- 3 d)
  Assess the testing coverage (proportion of patients with a result for each of the tests) to inform the feasibility of doing the tests proposed in this study for the assessment of the response to the use of two doses of amikacin
AE likely or definitely related to amikacin | at the end of treatment week 2 (+/- 3 d)
  Describe the occurrence of adverse events that are considered as likely or definitely related to the use of amikacin
amikacin concentration | during the first two treatment weeks
  Describe the amikacin concentration stratified by values for different treatment response markers : Colony forming units on semi-quantitative culture
amikacin concentration | during the first two treatment weeks
  Describe the amikacin concentration stratified by values for different treatment response markers : molecular bacterial load
amikacin concentration | during the first two treatment weeks
  Describe the amikacin concentration stratified by values for different treatment response markers : thin-layer agar semi-quantitative culture
amikacin concentration | during the first two treatment weeks
  Describe the amikacin concentration stratified by values for different treatment response markers: RNA Synthesis ratio
amikacin concentration | during the first two treatment weeks
  Describe the amikacin concentration stratified by values for different treatment response markers : time to culture positivity on liquid culture
post-injection pain | at 0, 15 minutes, 30 minutes and 60 minutes after the injection of amikacin with lidocaine on day 1 and 4, as well as the next morning
  Describe post-injection pain on a 0-10 pain scale (The Wong-Baker FACES pain rating scale) (15)
all AE, relationship with TB drugs | at the end of the ShORRT study, approximately 23 months after the treatment
  Describe all AE, by their grade, and their relationship with TB drugs
treatment outcomes | at the end of treatment
  Describe treatment outcomes, using the following effectiveness endpoints:
  * Month of stable (without reversion) culture conversion
  * End-of-treatment outcomes (treatment failure, death during treatment, LTFU during treatment, cure, treatment completion)
  * Treatment outcomes at 12 months post-treatment (end-of treatment outcome corrected for relapse)
  * Acquired resistance to bedaquiline, fluoroquinolone, amikacin through target deep sequencing on paired baseline and failure sputa
post-treatment outcomes | after post-treatment follow-up (part of ShORRT analysis)
  Describe post-treatment outcomes, using the following effectiveness endpoints:
  * Month of stable (without reversion) culture conversion
  * End-of-treatment outcomes (treatment failure, death during treatment, LTFU during treatment, cure, treatment completion)
  * Treatment outcomes at 12 months post-treatment (end-of treatment outcome corrected for relapse)
  * Acquired resistance to bedaquiline, fluoroquinolone, amikacin through target deep sequencing on paired baseline and failure sputa

CONTACTS AND LOCATIONS:
Overall Officials: Yves Habimana-Mucyo, MSc, Principal Investigator — Rwanda Biomedical Centre
Locations (1):
- Kabutare hospital, Kabutare, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snobre J, Gasana J, Ngabonziza JCS, Cuella-Martin I, Rigouts L, Jacobs BK, de Viron E, Herssens N, Ntihumby JB, Klibazayre A, Ndayishimiye C, Van Deun A, Affolabi D, Merle CS, Muvunyi C, Sturkenboom MGG, Migambi P, de Jong BC, Mucyo Y, Decroo T. Safety of high-dose amikacin in the first week of all-oral rifampicin-resistant tuberculosis treatment for the prevention of acquired resistance (STAKE): protocol for a single-arm clinical trial. BMJ Open. 2024 Jul 24;14(7):e078379. doi: 10.1136/bmjopen-2023-078379. PMID 39053960